CLINICAL TRIAL: NCT01818440
Title: Prospective Randomized Trial Comparing Navigation With 3D Roadmap vs. Conventional Angiography During Transarterial Embolization
Brief Title: Fluoroscopy or 3-D Roadmap Imaging Software for Liver Tumor Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 130092; 13-CC-0092
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08-22

CONDITIONS: Image-Guided Surgery
Keywords: Surgical Navigation; Liver; Cancer; Image-guided Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Patients will have the procedure performed with regular fluoroscopy (X-ray). Regular fluoroscopy is the standard method
  Interventions: Other: Fluoroscopy
- B (Experimental): Patients will have the procedure performed using the 3-D Roadmap software.With the 3DRoadmap, images from a Cone-Beam CT are analyzed. Software shows the vessels supplying the tumor and the plan is displayed on top of fluoroscopy
  Interventions: Other: 3D Roadmap software

INTERVENTIONS:
Other: 3D Roadmap software — Two scanning methods will be used by doctors to position catheters in the blood vessels to deliver the chemotherapy and close the blood supply to the tumor.
  Arms: B
Other: Fluoroscopy — Patients will have the procedure performed with regular fluoroscopy (X-ray). Regular fluoroscopy is the standard method.
  Arms: A

SUMMARY:
Background:

- Researchers are interested in comparing two methods that doctors can use to position catheters in blood vessels. These methods are used to deliver chemotherapy and close the blood supply to a tumor. The methods are the standard method called fluoroscopy and a new way called 3-D Roadmap. The 3-D Roadmap software uses computed tomography (CT) images to help the doctor choose the best position for the catheter to get to the tumor. The computer shows the route on an x-ray screen in real time. This technique may help doctors position the catheter with less x-ray dye and in a shorter time. These methods will be compared in people who are having a procedure to destroy liver tumors. The procedure, called trans-arterial embolization, will deliver chemotherapy and destroy the tumor blood supply.

Objectives:

- To compare the effectiveness of fluoroscopy or 3-D Roadmap software for liver tumor treatment.

Eligibility:

- Individuals at least 18 years of age who are having trans-arterial embolization for liver cancer.

Design:

* Participants will be screened with a physical exam and medical history. They will provide blood and urine samples, and have imaging studies.
* Participants will be divided into two groups. One group will have regular fluoroscopy (X-ray) during the procedure. The other group will have the procedure with the 3-D Roadmap software.
* In the first group, participants will have a CT scan. The doctor will decide how many vessels need to be treated. The doctor will advance the catheter using fluoroscopy only. Another CT scan will be given after the procedure.
* In the second group, participants will have a CT scan. The doctor will look at the scan with the 3-D Roadmap software. The software will show the path to advance the catheter. The doctor will use the software to help destroy the tumors. Another CT scan will be given after the procedure.
* Both groups will have the same follow-up care afterward. Other tests will be given as needed for the cancer treatment.

DETAILED DESCRIPTION:
Background:

This is a phase II prospective randomized trial comparing novel tumor segmentation and navigation with 3D roadmap vs. conventional imaging with angiography during trans-arterial embolization procedures. Cone beam CT (CBCT) obtains CT-like images in the angiography suite during trans-arterial chemoembolization procedures and liver chemo-perfusion (PHP). In addition, 2D liver perfusion metrics can be calculated from angiography images. 3D Roadmap is a navigation tool/ software that utilize the data from the CBCT overlaid on live fluoroscopy to display a segmented tumor, delineate its vascular supply and to navigate catheters to the target vessels. Moreover, with 3D Roadmap, CBCT can be fused to prior CT or MRI for improved target visualization. The 3D Roadmap software received 510 (k) clearance on February 19, 2004. Our CRADA partner, Philips Healthcare, also submitted and received a separate 510 (k) clearance on January 30, 2015 for the software s vessel segmentation functionality and is under the trade name Emboguide. 3D Roadmap/ Emboguide software is intended to be used in combination with the AlluraClarity X-ray system.

Primary Objective:

To compare safety, and technical efficiency of navigation with 3D Roadmap vs. conventional image guidance during trans-arterial embolization procedures.

Eligibility:

Subjects are eligible if:

* They are more than 18 years of age
* They have primary or metastatic hepatic tumors scheduled for trans-arterial chemo- embolization or bland embolization in interventional radiology
* They are eligible for trans-arterial chemoembolization or bland embolization

Subjects are excluded if they have:

* An altered mental status precluding understanding or consenting for the procedure
* Contra-indications to trans-arterial embolization
* A gross body weight exceeding 375 pounds (upper limit of angio table)
* A pregnancy
* A severe allergic reaction to iodine contrast which cannot be controlled by premedication with antihistamines and steroids

Design:

* Number of Participants: 30
* Recruitment Time Frame: 2 years
* Number of sites: 1
* Type of Study: prospective randomized clinical trial

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have primary or metastatic hepatic tumors scheduled for trans-arterial chemo-embolization or bland embolization in interventional radiology. A multi-disciplinary team including oncology, surgery, pathology and radiation oncology as well as interventional radiology will review each candidate and determine the eligibility for TACE or bland embolization and ineligibility for other interventions.
  2. Age >18 years
  3. They must be eligible for trans-arterial chemoembolization or bland embolization

EXCLUSION CRITERIA:

1. Patients with an altered mental status precluding understanding or consenting for the procedure
2. History of allergic reactions to iodine contrast, which cannot be controlled by premedication with antihistamines and steroids.
3. Pregnant women are excluded from the study because ionizing radiation is teratogenic or abortifacient effects. Patients are excluded from pregnancy testing if they are above the childbearing age of 55 years old, or if they have documented history of infertility or acquired or congenital disorders incompatible with pregnancy or if the patient has had a hysterectomy or bilateral oophorectomy. Patients are also excluded from pregnancy testing if they are at least 50 years of age AND have not menstruated for at least 12 months OR have a documented Follicle Stimulating Hormone (FSH) level of greater than 40 mIU/mL.
4. Patients with a total body weight exceeding 375 pounds since that is the weight limit of the angiography table.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-03-21; Primary Completion 2015-09-16 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
To compare safety, efficacy, and technical efficiency of navigation with 3D Roadmap vs. conventional image guidance during trans-arterial embolization procedures. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bradford J Wood, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Meyer BC, Witschel M, Frericks BB, Voges M, Hopfenmuller W, Wolf KJ, Wacker FK. The value of combined soft-tissue and vessel visualisation before transarterial chemoembolisation of the liver using C-arm computed tomography. Eur Radiol. 2009 Sep;19(9):2302-9. doi: 10.1007/s00330-009-1410-x. Epub 2009 May 8. PMID 19424701
- [Background] Li C, Heidt DG, Dalerba P, Burant CF, Zhang L, Adsay V, Wicha M, Clarke MF, Simeone DM. Identification of pancreatic cancer stem cells. Cancer Res. 2007 Feb 1;67(3):1030-7. doi: 10.1158/0008-5472.CAN-06-2030. PMID 17283135
- [Background] Wallace MJ, Murthy R, Kamat PP, Moore T, Rao SH, Ensor J, Gupta S, Ahrar K, Madoff DC, McRae SE, Hicks ME. Impact of C-arm CT on hepatic arterial interventions for hepatic malignancies. J Vasc Interv Radiol. 2007 Dec;18(12):1500-7. doi: 10.1016/j.jvir.2007.07.021. PMID 18057284